CLINICAL TRIAL: NCT06648798
Title: LIMBER UniLeg: Rapid, On-demand, and Scaled-up Manufacturing of Customized Transtibial Prosthetic Legs for Amputees
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LIMBER Prosthetics & Orthotics Inc (Industry)
Collaborators: University of California, San Diego (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 803632; 1R43HD112285-01A1 (NIH)
Record Dates: First submitted 2024-10-11; First posted 2024-10-18 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Amputation of Lower Limb; Prosthesis; Non-inferiority Trial of Prothesis
Keywords: Prosthesis; Trans-tibial amputation; Limber Unileg; 3D Printed

STUDY DESIGN:
Intervention Model Description: One study group of 30 participants involved for two months using a non-inferiority design in which the participant will be assessed using their normal device (1 month) and the study device (1 month).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will be involved for two months using a non-inferiority design in which the participant will be assessed using their normal device (1 month) and the study device (1 month).
  Interventions: Device: Limber Limb

INTERVENTIONS:
Device: Limber Limb — Participants will be involved for two months using a non-inferiority design in which the participant will be assessed using their normal device (1 month) and the study device (1 month).

SUMMARY:
The LIMBER UniLeg, a 3D printed single-piece transtibial prosthetic limb, is sufficiently equivalent to traditional passive prosthetic limbs (no motors or sensors), while reducing the cost and time of manufacturing and enabling global reach through the use of digital technologies to solve the worldwide prosthetic accessibility crisis. This is a single-site, Phase I, Clinical Research Study to test the effectiveness and safety of the LIMBER UniLeg. One study group of 30 participants involved for two months using a non-inferiority design in which the participant will be assessed using their normal device (1 month) and the study device (1 month).

DETAILED DESCRIPTION:
Globally, 35-40 million people need prosthetics or other assistive devices, and this number is expected to double by 2050 due to factors including an aging population and the rise in diabetes. However, only 5-15% of people in need have access to prosthetics or other assistive devices, in both underserved and developed countries. The result is that millions of people are denied basic quality of life because they can't walk, take care of themselves, or participate in society. The lack of availability stems from several factors including poor access to clinics and high cost. Prosthetic devices are hand-sculpted and assembled by prosthetists via complex and time-consuming processes. High-cost 3rd party components are used to connect and align the hand-crafted components, leading to an expensive end-product.

Currently, several companies are successfully delivering 3D printed prosthetic sockets, but no one can deliver a fully 3D printed, single piece 'unibody' prosthesis. 3D printed sockets have been shown to provide increased comfort and fit and streamline the manufacturing process, but using traditional pylon, ankle/foot, and connector components lead to many of the same issues as traditional devices. Only 3D printing the socket may improve the outcome for people who could have gotten a traditional device but leaves behind the people in need who don't have access in the first place.

The custom-fit requirements make it difficult to mass-produce affordable devices and a lack of access to proper health care and medical professionals prevents adjustments needed to maintain safe, comfortable, and reliable prosthetic devices. This is critically important during the early recovery period when residual limbs change in shape due to atrophy and scar tissue formation, as well as having nerve endings that may be extra- sensitive. For children who grow quickly and need new devices every few months or years, swift access is both physically and psychologically important. Small imperfections at the prosthesis-limb interface can cause severe discomfort and may be the difference between an amputee wearing their prosthesis or choosing to forgo mobility. To obtain a well-fitted socket, prosthetists take measurements of the residual limb with a fitted liner and then mark anatomical areas on the limb. After assessing the limb, the prosthetist will use plaster bandages to create a cast around the limb. The anatomical marks will transfer to the interior of the mold, such that the prosthetist can attempt to design the socket to consider regions of bone or soft tissue. The prosthetist can manipulate the plaster bandages while they are hardening to adjust its shape. This shaping requires years of experience and will only result in a comfortable, functional socket if the prosthetist is highly skilled. Due to the expensive and time-consuming nature of this traditional process, new solutions are urgently needed.

Clinical Trial Justification:

During this study the study team expects to gather both quantitative and qualitative data that will be used to produce a performance report on the functionality of the LIMBER UniLeg. The goal of this trial is to provide evidence of non-inferiority of the intervention compared to the functional performance of similarly featured passive prosthetic devices, e.g. the patient's existing device.

This clinical trial will quantify the functionality, clinical efficacy, and quality of care of the LIMBER UniLeg and compare it to traditional passive prosthetic devices, referred to as existing prosthetic devices (EPD). This will provide evidence that LIMBER's novel 3D printing, scanning, and digital design workflow produces devices that are not inferior to traditionally manufactured prosthetic limbs.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Persons, aged 18 to 75
4. In good general health as determined by clinical site monitor
5. Weight < 125kg
6. Are not diabetic (self reported)
7. Be a unilateral transtibial amputee of more than 1 year since amputation
8. Have an existing prosthetic device(s) that does not use sensors or motors (is passive)
9. Live in the Southern California region (within 50 miles of UCSD)
10. Has sufficient sensation in residual limb as tested by the clinical site monitor
11. Agreement to adhere to Lifestyle Considerations throughout study duration 11a. Use the testing device (EPD or UniLeg) only during the testing periods. 11b. Walk at least 14,000 steps per week (average of 1 mile per day). 11c. Maintain a similar diet and activity level throughout study duration (no abrupt changes of weight, activity, etc.)

Exclusion Criteria:

1. Not currently using a prosthetic device
2. Prosthetic device with active motors, sensors, etc.
3. Pregnancy (due to fall risk)
4. Diabetic (due to poor limb sensation), self reported
5. No under 18 (due to inability to consent)
6. No over 75 (due to fall risk)
7. Poor proprioception or sensation at the residual limb

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Mobility - 6min walk | Baseline, 4weeks, 8 weeks
  Measure total distance for a timed six-min walk test for both the Limber UniLeg vs. existing prosthetic devices.
Mobility - Timed-Up-and-Go | Baseline, 4weeks, 8 weeks
  Measure time for the timed up and go (TUG) test for both the Limber UniLeg vs. existing prosthetic devices.
Mobility--25 foot walk | All visits (Baseline, 4 weeks, 8 weeks)
  Time to cover 25 feet walking at a normal speed

SECONDARY OUTCOMES:
Quality of Care - Gait Symmetry | Baseline, 4weeks, 8 weeks
  Measure load distribution and stride length using a six-foot force pad test for both the UniLeg and existing prosthetic device to quantify gait symmetry.
Quality of Care - Perceived Balance Confidence_Limits of Stability | Baseline, 4weeks, 8 weeks
  Assess Participant's Limit of Stability using the NeuroCom Balance Manager. Metrics include movement velocity, directional control, and maximal excursion in 8 directions (cardinal and semi-cardinal). Higher scores are better and indicative of both a wider cone of stability (associated with less fall risk) and balance confidence (associated with greater overall movement and less fall rsik)
Quality of Care - Perceived Balance Confidence_Adaptation Test | Baseline, 4weeks, 8 weeks
  Assess Participant's Adaptation using the NeuroCom Balance Manager. Metrics include recovery time following a pertubation. Unit of measurement is milliseconds with higher scores being indicative of slower recovery (associated with higher fall risk). Across 5 trials participants are expected to improve.
  The degree of improvement (Score 1-Score 5) is also a metric of interest with higher scores associated with less fall risk.
Quality of Care - Perceived Balance Confidence_Motor Control | Baseline, 4weeks, 8 weeks
  Assess Participant's Motor Control using the NeuroCom Balance Manager. Metrics include stability following a pertubation. Unit of measurement is milliseconds with higher scores being indicative of slower recovery (associated with higher fall risk). Scores are averaged across multiple moderate and large pertubations in both the forward and backward directions.
Quality of Care - Utilization--At-home movement | Baseline-4weeks, 4weeks-8weeks
  Measure total steps measured for two weeks per assessment period using an Actigraph accelerometer. This will quantify utilization/daily ambulation while wearing the device(s), which will directly relate to patient satisfaction and comfort.
Quality of Care - Utilization--Physical Activity Intensity | Baseline-4weeks, 4weeks-8weeks
  Measure daily minutes spent in sedentary, light moderate, and intense levels of physical activity for two weeks per assessment period using an Actigraph accelerometer. This will quantify intensity of activity while wearing the device(s) which will directly relate to patient satisfaction and comfort, and effect on daily activity which may have impacts on other health metrics.
  Data will be derived based on movement levels using multiple potential cutpoints to quantify each minute as being one of the four potential activity bins. These are then summed across a day for activity level. Sleep time is removed by asking participants not to wear the device while in bed.

OTHER OUTCOMES:
Clinical Outcome - Pain | Baseline, 4weeks, 8 weeks
  Collect Numeric Pain Rating Scale (NPRS) measures for the UniLeg and existing prosthetic device to characterize the reduction in joint, lower back, and limb pain.
  The scale is completed on a visual slider and then measured by location to be between 1-100 with higher numbers being indicative of less pain/greater comfort.
Clinical Outcome - Quality of Life-European Quality of Life 5-Dimension 5-Level questionnaire | Baseline, 4weeks, 8 weeks
  Collect the European Quality of Life 5-Dimension 5-Level questionnaire (EQ5D5L) measures for the UniLeg and existing prosthetic device to characterize the improvements in health-related quality of life. The questionnaire is self-completed to assess five dimensions of health: Mobility, Self-care, Usual activities, Pain and discomfort, and Anxiety and depression on a 5 point scale from 1 (none) to 5 (extreme) with 5 being positive on mobility, self-care and usual activities and 1 on pain and anxiety subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Herb Barrack, CPO, Principal Investigator — LIMBER Prosthetics & Orthotics Inc
Locations (2):
- United States (2):
  - University of California San Diego, La Jolla, California
  - Limber Prosthetics & Orthotics Inc, San Diego, California

IPD SHARING:
Plan to Share IPD: No
Demographic and baseline outcomes will be presented using summary statistics. No individual data will be provided.

REFERENCES:
- [Background] Holm, S. A simple sequentially rejective multiple test procedure. Scandinavian journal of statistics, 6(2):65-70, 1979.
- [Background] Efron, B. and Tibshirani, R.J. An Introduction to the Bootstrap, Springer, New York, NY, 1993.
- [Background] US Department of Health and Human Services C for DC and P. Assessment Timed Up and Go (TUG).; 2017. Accessed June 12, 2018
- [Background] Sions JM, Beisheim EH, Manal TJ, Smith SC, Horne JR, Sarlo FB. Differences in Physical Performance Measures Among Patients With Unilateral Lower-Limb Amputations Classified as Functional Level K3 Versus K4. Arch Phys Med Rehabil. 2018 Jul;99(7):1333-1341. doi: 10.1016/j.apmr.2017.12.033. Epub 2018 Feb 1. PMID 29410114
- [Background] Reid L, Thomson P, Besemann M, Dudek N. Going places: Does the two-minute walk test predict the six-minute walk test in lower extremity amputees? J Rehabil Med. 2015 Mar;47(3):256-61. doi: 10.2340/16501977-1916. PMID 25588644
- [Background] Dite W, Connor HJ, Curtis HC. Clinical identification of multiple fall risk early after unilateral transtibial amputation. Arch Phys Med Rehabil. 2007 Jan;88(1):109-14. doi: 10.1016/j.apmr.2006.10.015. PMID 17207685
- [Background] McCaffrey M, Beebe A. Managing your patients' adverse reactions to narcotics. Nursing. 1989 Oct;19(10):166-8. No abstract available. PMID 2586868
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Heil DP, Brage S, Rothney MP. Modeling physical activity outcomes from wearable monitors. Med Sci Sports Exerc. 2012 Jan;44(1 Suppl 1):S50-60. doi: 10.1249/MSS.0b013e3182399dcc. PMID 22157775
- [Background] Bassett DR Jr, Rowlands A, Trost SG. Calibration and validation of wearable monitors. Med Sci Sports Exerc. 2012 Jan;44(1 Suppl 1):S32-8. doi: 10.1249/MSS.0b013e3182399cf7. PMID 22157772
- [Background] Freedson P, Bowles HR, Troiano R, Haskell W. Assessment of physical activity using wearable monitors: recommendations for monitor calibration and use in the field. Med Sci Sports Exerc. 2012 Jan;44(1 Suppl 1):S1-4. doi: 10.1249/MSS.0b013e3182399b7e. PMID 22157769
- [Background] Rostagno C, Gensini GF. Six minute walk test: a simple and useful test to evaluate functional capacity in patients with heart failure. Intern Emerg Med. 2008 Sep;3(3):205-12. doi: 10.1007/s11739-008-0130-6. Epub 2008 Feb 26. PMID 18299800
- [Background] Solway S, Brooks D, Lacasse Y, Thomas S. A qualitative systematic overview of the measurement properties of functional walk tests used in the cardiorespiratory domain. Chest. 2001 Jan;119(1):256-70. doi: 10.1378/chest.119.1.256. PMID 11157613
- [Background] Bartels B, de Groot JF, Terwee CB. The six-minute walk test in chronic pediatric conditions: a systematic review of measurement properties. Phys Ther. 2013 Apr;93(4):529-41. doi: 10.2522/ptj.20120210. Epub 2012 Nov 15. PMID 23162042
- [Background] Bui KL, Nyberg A, Maltais F, Saey D. Functional Tests in Chronic Obstructive Pulmonary Disease, Part 1: Clinical Relevance and Links to the International Classification of Functioning, Disability, and Health. Ann Am Thorac Soc. 2017 May;14(5):778-784. doi: 10.1513/AnnalsATS.201609-733AS. PMID 28244799
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Sprint G, Cook DJ, Weeks DL. Toward Automating Clinical Assessments: A Survey of the Timed Up and Go. IEEE Rev Biomed Eng. 2015;8:64-77. doi: 10.1109/RBME.2015.2390646. Epub 2015 Jan 12. PMID 25594979
- [Background] Barry E, Galvin R, Keogh C, Horgan F, Fahey T. Is the Timed Up and Go test a useful predictor of risk of falls in community dwelling older adults: a systematic review and meta-analysis. BMC Geriatr. 2014 Feb 1;14:14. doi: 10.1186/1471-2318-14-14. PMID 24484314
- [Background] Schoene D, Wu SM, Mikolaizak AS, Menant JC, Smith ST, Delbaere K, Lord SR. Discriminative ability and predictive validity of the timed up and go test in identifying older people who fall: systematic review and meta-analysis. J Am Geriatr Soc. 2013 Feb;61(2):202-8. doi: 10.1111/jgs.12106. Epub 2013 Jan 25. PMID 23350947
- See also: Limber Prosthetics Website — https://www.limberprosthetics.com/